CLINICAL TRIAL: NCT04972487
Title: Global Early Access Program to Provide Tofersen To Patients With Amyotrophic Lateral Sclerosis (ALS) Associated With a Mutation in the Superoxide Dismutase 1 (SOD1) Gene
Brief Title: Expanded Access Program for Tofersen in Participants With Superoxide Dismutase 1-Amyotropic Lateral Sclerosis
Status: Approved for marketing | Type: Expanded Access
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 233AS001
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Superoxide Dismutase 1-Amyotropic Lateral Sclerosis
MeSH Terms: interventions — tofersen

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Tofersen — Administered as intrathecal bolus injection
  Other Names: BIIB067; QALSODY

SUMMARY:
The objective of this early access program (EAP) is to provide access to tofersen to eligible participants with amyotrophic lateral sclerosis (ALS) associated with a mutation in the superoxide dismutase 1 (SOD1) gene prior to an alternative access mechanism in order to address a high unmet medical need in this population.

DETAILED DESCRIPTION:
Treating healthcare professionals (HCPs) of participants who meet the inclusion/exclusion criteria may request access by emailing medicineaccess@clinigengroup.com. The current EAP structure does not limit participants to receive access at specific sites. Treating HCPs can submit requests on behalf of participants by emailing Clinigen at the email address provided below. Information on the EAP eligibility criteria, including participants and center criteria, will be provided by Clinigen as part of the enrollment request process.

ELIGIBILITY:
Key Inclusion Criteria:

* Medically able to undergo the program procedures, as determined by the treating healthcare professional (HCP).
* Weakness attributable to ALS and associated with a mutation in the SOD1 gene (SOD1-ALS).

Key Exclusion Criteria:

* Previous or current participation in a clinical trial of tofersen.
* Use of an investigational medicinal product (IMP) for amyotrophic lateral sclerosis (ALS) within 5 half-lives of the IMP before the first dose of tofersen.
* Participant's primary place of residence is outside of the country of treatment.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (19):
- United States (19):
  - Research Site, Anchorage, Alaska
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Chicago, Illinois
  - Research Site, Kansas City, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lebanon, New Hampshire
  - Research Site, Amherst, New York
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas